CLINICAL TRIAL: NCT03460665
Title: Symptomatic Efficacy of Microparticle Arterial Embolization in Knee Osteoarthritis Resistant to Medical Treatment: Randomized Prospective Study Versus Placebo
Brief Title: Symptomatic Efficacy of Microparticle Arterial Embolization in Knee Osteoarthritis Resistant to Medical Treatment
Acronym: EMBARGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-PP-01
Record Dates: First submitted 2018-02-06; First posted 2018-03-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microparticles (Experimental): arteriography and an injection of inert microparticles of 75 µm in neovessels
  Interventions: Procedure: Arteriography
- Placebo (Placebo Comparator): knee arteriography and injection of saline solution in neovessels
  Interventions: Procedure: Arteriography

INTERVENTIONS:
Procedure: Arteriography — knee arteriography

SUMMARY:
The aim of this double-blind, randomized, single-center prospective study (patient and evaluator) is to evaluate the efficacy of arterial occlusion (embolization) of neovessels by microparticle versus placebo on pain in disabling knee osteoarthritis at 12 months.

DETAILED DESCRIPTION:
Rational: in the normal state, the articular cartilage is devoid of vessels and innervation. In osteoarthritic cartilage, neovascularization is observed and is accompanied by a sensitive neoinnervation. The development of these neovessels also contributes to the structural damage of cartilage by achieving a real "perforation"of the cartilage. Studies designate neovascularization as a target for new therapeutic. In two non-comparative open-label studies, a Japanese team has shown that endovascular occlusion of these neovessels in patients with knee osteoarthritis significantly reduced the patient pain without any complication.

The aim of this double-blind, randomized, single-center prospective study (patient and evaluator) is to evaluate the efficacy of arterial occlusion (embolization) of neovessels by microparticle versus placebo on pain in disabling knee osteoarthritis at 12 months.

The main objective is to evaluate the effectiveness of embolization on the pain of patients with disabling osteoarthritis by double-blind comparison of two groups: the first control group will include patients who will benefit from arteriography and an injection of saline in their neovessels, the second group called treatment will consist of patients whose neovessels will be occluded by inert microparticles of 75 µm. The pain will be evaluated in both groups before and 12 months after embolisation. The objective is to show that the pain is significantly less important in the group of patients whose neovessels have been occluded with microparticles in comparison to the control group.

Secondary objectives are to evaluate the effectiveness of neovascular embolization on pain at 1, 6, 24 and 36 months; knee stiffness, physical activity, quality of life, at 1, 6, 12, 24 and 36 months; the structural course of knee osteoarthritis at 12, 24 and 36 months; the use of arthroplasty at 24 and 36 months.

Study Population: Patients aged 40 to 80 years with knee osteoarthritis with a visual analogue scale (VAS) score greater than or equal to 50 mm for at least 3 months optimal medical treatment, whose radiological stage of osteoarthritis according to Kellgren and Lawence is 2 or 3 and does not have a knee prosthesis surgical indication.

Primary endpoint: modification of the pain item of the self-administered Knee injury and Osteoarthritis Outcome Score (KOOS) collected in the 15 days preceding the procedure and at 12 months.

Secondary evaluation criteria are KOOS, EQ-5D (Quality of Life Scale) in the 15 days preceding the procedure and then at 1, 6, 24 and 36 months; knee radiographs, number of patients who had 12, 24 and 36 months of joint replacement surgery; knee MRI at 12 months; the use of analgesics and anti-inflammatories; adverse events.

Expected benefits: confirm the results of the non-randomized studies that showed a clear decrease in pain related to knee osteoarthritis after occlusion of neovessels, allowing the reduction of antalgic drug consumption, improving the quality of life of patients of this pathology, delay the need for prosthetic surgery.

ELIGIBILITY:
Inclusion Criteria:

* An effective contraceptive system for women of childbearing age, a pregnancy test will be offered to these women in the preoperative assessment.
* Obtaining the signature of the consent to participate in the study
* Kellgren-Lawrence (KL) grade 2-3 assessed by routine weight-bearing knee radiographs on the most affected knee in bilateral cases
* Pain with EVA ≥ 50 mm evolving for at least 3 months despite the start of a well-conducted medical treatment according to current recommendations including analgesics, NSAID, intra-articular injections, rehabilitation and weight loss
* No surgical indication retained

Exclusion Criteria:

* Serious visceral failure
* Local infection
* Arthropathy secondary to chronic inflammatory rheumatism (rheumatoid arthritis, spondylarthritis) or microcrystalline rheumatism
* History of surgery on the studied knee, except arthroscopy for more than 6 months
* Gonarthrosis with KL score> 3
* Osteonecrosis of one of the bones of the knee joint on the MRI
* Pregnant or lactating woman
* Allergy to contrast products
* Chronic or acute renal failure (clearance <30 ml / min)
* Haemostasis disorders (blood platelet count <50,000 / mm3 or patient ACT / control ACT> 1,2 or PT <50%)
* Operative indication of placement of a prosthesis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
VAS : Change of pain of the Knee injury | before intervention and one month, 6 months, 12 months, 24 months and 36 months after intervention
  change in the Visual Analog Scale of Pain Intensity (VASPI).

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | at 1,6, 24, 36 month after intervention
  KOOS questionnaire assess changes from month to month induced by treatment. KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale
EQ-5D questionnaire | at 1, 6, 12 and 36 month after intervention
  EQ-5D questionnaire is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale.
Knee MRI | 15 days before embolization and 12 month after
  Knee MRI
Knee X-Ray | 15 days before embolization and 12, 24, 36 month after
  Knee X-Ray

CONTACTS AND LOCATIONS:
Overall Officials: Yves CHAU HUU DANH, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - chu Bordeaux, Bordeaux
  - BREUIL, Nice
  - Chu de Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No